CLINICAL TRIAL: NCT06592079
Title: Hard and Soft Tissue Changes After Immediate Implant Placement Using Connective Tissue Graft With and Without Bone Grafting in the Esthetic Zone: A Randomized Clinical Trial
Brief Title: Hard and Soft Tissue Changes After Immediate Implant Placement Using Connective Tissue Graft With and Without Bone Grafting in the Esthetic Zone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norai Ahmed Mohamed Zayed, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 924
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Immediate Implants Connective Tissue Graft
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant & Connective tissue graft (Experimental): Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supra-periosteal partial dissection pouch prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place. Followed by customized healing abutment.
  Interventions: Procedure: Immediate implant and connective tissue graft
- Immediate implant with connective tissue graft & bone graft (Active Comparator): Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supra-periosteal partial dissection pouch prepared at the buccal aspect without using vertical incisions and without flap elevation. Xenograft will be used to fill the jumping gap.Sutures will be used to stabilize the graft in its desired place. Followed by customized healing abutment.
  Interventions: Procedure: Immediate implant with connective tissue graft and bone graft

INTERVENTIONS:
Procedure: Immediate implant and connective tissue graft — Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supra-periosteal partial dissection pouch prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place. Followed by customized healing abutment.
  Arms: Immediate implant & Connective tissue graft
Procedure: Immediate implant with connective tissue graft and bone graft — Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supra-periosteal partial dissection pouch prepared at the buccal aspect without using vertical incisions and without flap elevation. Xenograft will placed to fill the jumping gap.Sutures will be used to stabilize the graft in its desired place. Followed by customized healing abutment.
  Arms: Immediate implant with connective tissue graft & bone graft

SUMMARY:
Evaluation of soft and hard tissue changes after immediate implant placement with connective tissue graft and bone as a control group and connective tissue graft only as a test group.

DETAILED DESCRIPTION:
This randomized clinical trial will evaluate the effect of using connective tissue graft and bone graft versus connective tissue graft, with customized healing abutments during immediate implant placement on volumetric mid facial recession .In patients with type I socket who need extraction in the anterior maxilla.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:
* Adults at or above the age of 18.
* Non-restorable maxillary anterior or premolar tooth requiring extraction and needed an implant placing therapy.
* The failing tooth will have adjacent and opposing natural teeth.
* Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration.
* Able to tolerate surgical periodontal procedures.
* Full mouth plaque and bleeding scores less than 20%.
* Compliance with the maintenance program.
* Provide informed consent.
* Accepts the one-year follow-up period.

Teeth related criteria:

* Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
* Intact socket wall before the extraction, buccal bone thickness ≤1mm assessed by CBCT.
* Sufficient apical bone to place an immediate implant with minimum primary stability of 30Ncm

Exclusion Criteria:

* Patients diagnosed with periodontal diseases.
* Current or previous smokers.
* Pregnant and lactating females.
* Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking IV Bis-phosphonates for treatment of osteoporosis.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with parafunctional habits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Volumetric Analysis of Mid-facial recession | Preoperative,3months,6months and 12 months
  3d viewer will be used to the the midfacial recession .

SECONDARY OUTCOMES:
Volumetric analysis of Interdental papillae height | Preoperative , 3 months, 6 months and 12 months
Bone formed labial to the implant | Preoperative and 1 year
Horizontal labio-palatal bone collapse | Preoperative and 1 year
Vertical crestal bone level changes | Preoperative and 1 year
Gingival biotype | Preoperative, 6 months and 12 months
Volumetric analysis of buccal contour | Preoperative,3months,6months and 12 months
Horizontal labio-palatal bone collapse | (Preoperative and 1 year)
Full mouth bleeding score (FMBS) | Preoperative, 6months and 12 months
  (0,1,2,3) 0:normal gingiva, 1: No bleeding , 2:bleeding on probing, 3:tendency to spontaneous bleeding.
Pain and discomfort | At 1,3 and 7 days after the surgery
  will be assessed using the visual analog scale VAS as recorded by the patient 1, 3 and 7 days after the surgery. The patients will mark the pain perception in a non-numerical 100 mm line ranging from "no pain=0" (left) to "very painful=100" (right). It will be given a numerical value by measuring in millimeters the distance from the left end of the line .
Full mouth plaque score (FMPS) | Preoperative, 6 months and 12 months
  0 : no plaque scored at gingival margin
  1: Plaque scored at gingival margin FMPS: Number of sites scored with plaque/Number of sites evaluated x 100
Pink Esthetic Score | at 12 months
  PES is based on seven parameters; mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color, and texture. The peri-implant mucosa will be evaluated by the seven index points.The contralateral tooth and the adjacent soft tissue served as reference using a 0-1-2 scoring system, with 0 being the lowest and 2 being the highest value.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year